CLINICAL TRIAL: NCT02095132
Title: A Phase 1/2 Study of AZD1775 (MK-1775) in Combination With Oral Irinotecan in Children, Adolescents, and Young Adults With Relapsed or Refractory Solid Tumors
Brief Title: Adavosertib and Irinotecan Hydrochloride in Treating Younger Patients With Relapsed or Refractory Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00547; NCI-2014-00547 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ADVL1312 (Other: Pediatric Early Phase Clinical Trial Network); ADVL1312 (Other: CTEP); UM1CA097452 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-03-24 (Estimated); Results first posted 2022-10-05 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-08

CONDITIONS: Central Nervous System Embryonal Tumor With Rhabdoid Features; Central Nervous System Embryonal Tumor, Not Otherwise Specified; Central Nervous System Ganglioneuroblastoma; Embryonal Tumor With Multilayered Rosettes, C19MC-Altered; Pineoblastoma; Primary Central Nervous System Neoplasm; Recurrent Childhood Central Nervous System Embryonal Neoplasm; Recurrent Malignant Solid Neoplasm; Recurrent Medulloblastoma; Recurrent Neuroblastoma; Recurrent Rhabdomyosarcoma; Refractory Malignant Solid Neoplasm; Refractory Medulloblastoma; Refractory Neuroblastoma; Refractory Rhabdomyosarcoma
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive; Pinealoma; Central Nervous System Neoplasms; Medulloblastoma; Neuroblastoma; Rhabdomyosarcoma | interventions — adavosertib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (irinotecan hydrochloride, adavosertib) (Experimental): Patients receive irinotecan hydrochloride PO and adavosertib PO on days 1-5. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Drug: Irinotecan Hydrochloride

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD-1775; AZD1775; MK-1775; MK1775
Drug: Irinotecan Hydrochloride — Given PO
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E

SUMMARY:
This phase I/II trial studies the side effects and best dose of adavosertib and irinotecan hydrochloride in treating younger patients with solid tumors that have come back (relapsed) or that have not responded to standard therapy (refractory). Adavosertib and irinotecan hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the maximum tolerated dose (MTD) and/or recommended phase 2 dose of adavosertib (AZD1755 [MK-1775]) administered on days 1 through 5 every 21 days, in combination with oral irinotecan (irinotecan hydrochloride), to children with recurrent or refractory solid tumors.

II. To define and describe the toxicities of AZD1755 (MK-1775) in combination with oral irinotecan administered on this schedule.

III. To characterize the pharmacokinetics of AZD1755 (MK-1775) in children with refractory cancer.

SECONDARY OBJECTIVES:

I. To preliminarily define the antitumor activity of AZD1755 (MK-1775) and irinotecan within the confines of a Phase 1 study.

II. To obtain initial phase 2 efficacy data on the anti-tumor activity of AZD1755 (MK-1775) in combination with irinotecan administered to children with relapsed or refractory neuroblastoma, in children with relapsed or refractory medulloblastoma/CNS PNET (central nervous system primitive neuroectodermal tumor) and in children with relapsed or refractory rhabdomyosarcoma.

III. To investigate checkpoint over-ride by AZD1755 (MK-1775) via the mechanism-based pharmacodynamic (PD) biomarker of decreased cyclin-dependent kinase 1 (CDK1) phosphorylation in correlative and exploratory studies.

IV. To evaluate potential predictive biomarkers of AZD1755 (MK-1775) sensitivity, including v-myc avian myelocytomatosis viral oncogene homolog (MYC), v-myc avian myelocytomatosis viral oncogene neuroblastoma derived homolog (MYCN), phosphorylated-WEE1 G2 checkpoint kinase (p-Wee1), enhancer of zeste homolog 2 (Drosophila) (EZH2) and gamma-H2A histone family, member gamma-(H2AX) in tumor tissues in correlative and exploratory studies.

OUTLINE: This is a phase I, dose-escalation followed by a phase II study.

Patients receive irinotecan hydrochloride orally (PO) and adavosertib PO on days 1-5. Treatment repeats every 21 days for up to 18 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG)
* Part A: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors
* Part B: Patients with relapsed or refractory neuroblastoma
* Part C: Patients with relapsed or refractory medulloblastoma or CNS embryonal tumors formally classified as PNET (pineoblastoma, CNS neuroblastoma, CNS ganglioneuroblastoma, embryonal tumor with multi-layered rosettes, medulloepithelioma, CNS embryonal tumor with rhabdoid features [INI1 intact] and CNS embryonal tumor, not otherwise specified)
* Part D: Patients with relapsed or refractory rhabdomyosarcoma
* Part A: Patients must have a body surface area >= 0.35 m^2 at the time of study enrollment if enrolling on dose levels 1-5; patients must have a body surface area >= 0.46 m^2 at the time of study enrollment if enrolling on dose level 0
* Parts B, C, and D: Phase 2 Expansion: Patients must have a body surface area of > 0.49 m^2 at the time of study enrollment at the recommended phase 2 dose of AZD-1775
* Part A: Patients must have either measurable or evaluable disease
* Part B: Patients must have either measurable disease or must be evaluable for MIBG response without evidence of Response Evaluation Criteria in Solid Tumors (RECIST) measurable lesions; patients with neuroblastoma in bone marrow only are not eligible
* Part C: Patients must have measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI)
* Part D: Patients must have measurable disease for Part D
* Patient's current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival with an acceptable quality of life
* Karnofsky >= 50% for patients > 16 years of age and Lansky >= 50 for patients =< 16 years of age; note: neurologic deficits in patients with CNS tumors must have been relatively stable for at least 7 days prior to study enrollment; patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score
* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy
* At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea)
* At least 14 days after the last dose of a long-acting growth factor (e.g. Neulasta) or 7 days for short-acting growth factor; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 7 days after the last dose of a biologic agent; for agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur; the duration of this interval must be discussed with the study chair
* At least 42 days after the completion of any type of immunotherapy, e.g. tumor vaccines
* >= 21 days must have elapsed from infusion of lase dose of antibody, and toxicity related to prior antibody therapy must be recovered to grade =< 1
* At least 14 days after local palliative radiation therapy (XRT) (small port); at least 150 days must have elapsed if prior traumatic brain injury (TBI), craniospinal XRT or if >= 50% radiation of pelvis; at least 42 days must have elapsed if other substantial bone marrow radiation, including therapeutic doses of iobenguane (MIBG)
* Stem cell Infusion without TBI: no evidence of active graft vs host disease and at least 84 days must have elapsed after transplant or stem cell infusion
* Patients previously treated with irinotecan are eligible for this study
* For patients with solid tumors without known bone marrow involvement: peripheral absolute neutrophil count (ANC) >= 1000/mm^3
* For patients with solid tumors without known bone marrow involvement: platelet count >= 100,000/mm^3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
* For patients with solid tumors without known bone marrow involvement: hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions)
* Patients with known bone marrow metastatic disease will be eligible for study provided they meet the blood counts (may receive transfusions provided they are not known to be refractory to red cell or platelet transfusions); these patients will not be evaluable for hematologic toxicity; at least 2 of every cohort of 3 patients must be evaluable for hematologic toxicity for Part A, the dose escalation part of the study; if dose-limiting hematologic toxicity is observed, all subsequent patients enrolled must be evaluable for hematologic toxicity
* Creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2 or a serum creatinine based on age/gender as follows:

  * Age 1 to < 2 years: 0.6 mg/dL
  * Age 2 to < 6 years: 0.8 mg/dL
  * Age 6 to < 10 years: 1 mg/dL
  * Age 10 to < 13 years: 1.2 mg/dL
  * Age 13 to < 16 years: 1.5 mg/dL (males), 1.4 mg/dL (females)
  * Age >= 16 years: 1.7 mg/dL (males), 1.4 mg/dL (females)
* Bilirubin (sum of conjugated + unconjugated) =< 1.5 x upper limit of normal (ULN) for age
* Serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 135 U/L; for the purpose of this study, the ULN for SGPT is 45 U/L
* Serum albumin >= 2 g/dL
* Correct QT interval (QTc) =< 480 msec; Note: Patients should avoid concomitant medication known or suspected to prolong QTc interval or cause torsades de pointes; if possible, alternative agents should be considered; patients who are receiving drugs that prolong the QTc are eligible if the drug is necessary and no alternatives are available
* Patients with seizure disorder may be enrolled if on non-enzyme inducing anticonvulsants and well controlled
* Nervous system disorders (Common Terminology Criteria for Adverse Events version 5.0 [CTCAE v5.0]) resulting from prior therapy must be =< grade 2, with the exception of decreased tendon reflex (DTR); any grade of DTR is eligible
* All patients and/or their parents or legally authorized representatives must sign a written informed consent; assent, when appropriate, will be obtained according to institutional guidelines
* Tissue blocks or slides must be sent if available, with exclusions; if tissue blocks or slides are unavailable, the study chair must be notified prior to study enrollment
* Patients must be able to swallow capsules

Exclusion Criteria:

* Pregnant or breast-feeding women may not be entered on this study as there is yet no available information regarding human fetal or teratogenic toxicities; pregnancy tests must be obtained in girls who are post-menarchal
* Males or females of reproductive potential may not participate unless they have agreed to use an effective double barrier contraceptive method for the entire duration of protocol therapy and for 3 months (males) and 1 month (females) after study drug discontinuation
* Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible
* Patients who are currently receiving another investigational drug are not eligible
* Patients who are currently receiving other anti-cancer agents are not eligible
* Patients who are currently receiving drugs that are strong or moderate inhibitors and/or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) or sensitive CYP3A4 substrates and CYP3A4 substrates with a narrow therapeutic range are not eligible; the use of aprepitant as an antiemetic is prohibited due to early drug interaction data demonstrating increased exposure to AZD1775 (MK-1775); caution should be exercised with concomitant administration of AZD1755 (MK-1775) and agents that are sensitive substrates of cytochrome P450, family 2, subfamily C, polypeptide 8 (CYP2C8), 2C9 and 2C19, or substrates of this enzyme with narrow therapeutic ranges, as well as agents that are inhibitors or substrates of permeability glycoprotein (P-gp)
* Patients who are receiving cyclosporine, tacrolimus or other agents to prevent graft-versus-host disease post bone marrow transplant are not eligible for this trial
* Patients must not have received enzyme inducing anticonvulsants for at least 14 days prior to enrollment
* Patients with cardiac diseases ongoing or in the past 6 months (e.g. congestive heart failure, acute myocardial infarction, significant uncontrolled arrhythmias) are not eligible for this trial
* Patients who have an uncontrolled infection are not eligible
* Patients who have received a prior solid organ transplantation are not eligible
* Patients who in the opinion of the investigator may not be able to comply with the safety monitoring requirements of the study are not eligible
* Patients with a history of allergic reaction to irinotecan, cephalosporins or a severe penicillin allergy are not eligible
* Patients unable to swallow capsules whole are not eligible; nasogastric or gastric (G) tube administration is not allowed

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina A Cole, Principal Investigator — COG Phase I Consortium
Locations (24):
- United States (23):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients must have had histologic verification of malignancy at original diagnosis or relapse except in patients with intrinsic brain stem tumors, optic pathway gliomas, or patients with pineal tumors and elevations of cerebrospinal fluid (CSF) or serum tumor markers including alpha-fetoprotein or beta-human chorionic gonadotropin (HCG).
Groups:
- Part A, Dose Level 1: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated at 70 mg/m2 Irinotecan (IRIN) and 50 mg/m2 AZD1775 (MK-1775)
- Part A, Dose Level 2: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated at 70 mg/m2 Irinotecan (IRIN) and 65 mg/m2 AZD1775 (MK-1775)
- Part A, Dose Level 3: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated at 90 mg/m2 Irinotecan (IRIN) and 65 mg/m2 AZD1775 (MK-1775)
- Part A, Dose Level 4: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated at 90 mg/m2 Irinotecan (IRIN) and 85 mg/m2 AZD1775 (MK-1775)
- Part A, Dose Level 5: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated at 90 mg/m2 Irinotecan (IRIN) and 110 mg/m2 AZD1775 (MK-1775)
- Part A, PK Expansion: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated at the MTD/RP2D of 90 mg/m2 Irinotecan (IRIN) and 110 mg/m2 AZD1775 (MK-1775)
- Part B, Neuroblastoma: Patients with relapsed or refractory neuroblastoma treated at the MTD/RP2D of 90 mg/m2 Irinotecan (IRIN) and 85 mg/m2 AZD1775 (MK-1775)
- Part C, Medulloblastoma/CNS PNET: Patients with relapsed or refractory Medulloblastoma/CNS PNET treated at the MTD/RP2D of 90 mg/m2 Irinotecan (IRIN) and 85 mg/m2 AZD1775 (MK-1775)
- Part D, Rhabdomyosarcoma: Patients with relapsed or refractory Rhabdomyosarcoma treated at the MTD/RP2D of 90 mg/m2 Irinotecan (IRIN) and 85 mg/m2 AZD1775 (MK-1775)
Period: Overall Study
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion | Part B, Neuroblastoma | Part C, Medulloblastoma/CNS PNET | Part D, Rhabdomyosarcoma
Started | 4 | 5 | 4 | 10 | 8 | 6 | 19 | 10 | 10
Completed | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Not Completed | 4 | 5 | 4 | 10 | 7 | 6 | 18 | 9 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 3 | 5 | 2 | 8 | 3 | 6 | 10 | 9 | 8
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 3 | 0 | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion | Part B, Neuroblastoma | Part C, Medulloblastoma/CNS PNET | Part D, Rhabdomyosarcoma | Total
Number analyzed (Participants) | 4 | 5 | 4 | 10 | 8 | 6 | 19 | 10 | 10 | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 4 | 7 | 6 | 4 | 18 | 8 | 10 | 64
  Between 18 and 65 years | 1 | 1 | 0 | 3 | 2 | 2 | 1 | 2 | 0 | 12
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Years] | 15 [10 to 19] | 16 [7 to 19] | 13.5 [11 to 15] | 11 [7 to 20] | 14.5 [5 to 20] | 10.5 [2 to 19] | 9 [6 to 19] | 13.5 [6 to 20] | 11 [4 to 16] | 11.5 [2 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 5 | 3 | 7 | 6 | 2 | 31
  Male | 2 | 3 | 2 | 8 | 3 | 3 | 12 | 4 | 8 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 2 | 8
  Not Hispanic or Latino | 3 | 5 | 4 | 9 | 6 | 6 | 16 | 9 | 7 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 1 | 0 | 2 | 4 | 3 | 0 | 10
  White | 4 | 4 | 1 | 8 | 5 | 4 | 11 | 7 | 9 | 53
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: MTD is defined as the maximum doses of adavosertib and irinotecan hydrochloride at which fewer than one-third of patients experience dose limiting toxicities when receiving this combination.
Time Frame: Up to 21 days
Population: All Part A patients contributed to determining MTD. Only Toxicity evaluable patients were accounted.
Measure: Number; unit: mg/m^2
Groups:
- Part A: Part A Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated with Irinotecan (IRIN) and AZD1775 (MK-1775)
Arm/Group | Part A
Number analyzed (Participants) | 27
mg/m^2
  Irinotecan (IRIN) | 90
  AZD1775 (MK-1775) | 85

2. Primary Outcome: Number of Participants With Cycle 1 DLT
Description: To define and describe the toxicities of AZD1755 (MK-1775) in combination with oral irinotecan administered on this schedule.
Time Frame: Up to 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion | Part B, Neuroblastoma | Part C, Medulloblastoma/CNS PNET | Part D, Rhabdomyosarcoma
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 6 | 6 | 16 | 7 | 7
Participants | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1

3. Primary Outcome: Pharmacokinetic (PK) Parameters of Adavosertib in Terms of Systemic Exposure, AUC
Description: The PK parameters will be summarized by means and standard deviations
Time Frame: Cycle 1 day 1 prior to the irinotecan infusion, prior to the adavosertib dose, 4 hours after the dose of adavosertib is given, and prior to the irinotecan dose on day 2
Population: Summary statistics for PK parameter for patients in Part A. Per study protocol, PK measures were not required for Parts B, C, or D, therefore, data were not and will not be collected.
Measure: Mean (Standard Deviation); unit: hr*nmol/L
Groups:
- Part A, Dose Level 1: Patients with relapsed or refractory solid tumors, including patients with primary or metastatic CNS tumors treated at 70 mg/m2 Irinotecan (IRIN) and 50 mg/m2 AZD1775 (MK-1775
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion
Number analyzed (Participants) | 4 | 4 | 4 | 8 | 5 | 4
hr*nmol/L | 3222.95 (1770.92) | 3397.3 (2404.13) | 4413.22 (2026.63) | 5344.96 (1839.62) | 5161.36 (3282.31) | 4655.13 (1943.68)

4. Primary Outcome: Pharmacokinetic (PK) Parameters of Adavosertib in Terms of Systemic Exposure, Cmax
Description: The PK parameters will be summarized by means and standard deviations
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion
Number analyzed (Participants) | 4 | 4 | 4 | 8 | 5 | 4
nmol/L | 443.96 (168.13) | 511.23 (341.4) | 539.84 (265.58) | 652.71 (240.27) | 733.59 (397.41) | 590.28 (378.65)

5. Primary Outcome: Pharmacokinetic (PK) Parameters of Adavosertib in Terms of Systemic Exposure, HL-Lambda (Half Life)
Description: The PK parameters will be summarized by means and standard deviations
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion
Number analyzed (Participants) | 4 | 4 | 4 | 8 | 5 | 4
hours | 4.7 (1) | 5.5 (3.9) | 5.7 (1.3) | 4.9 (1) | 4 (2.1) | 4.7 (0.6)

6. Primary Outcome: Pharmacokinetic (PK) Parameters of Adavosertib in Terms of Systemic Exposure, Tmax
Description: The PK parameters will be summarized by means and standard deviations
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion
Number analyzed (Participants) | 4 | 4 | 4 | 8 | 5 | 4
hours | 3.5 (3) | 2 (1.3) | 3 (1.1) | 3 (1.1) | 2.4 (0.9) | 3.5 (3)

7. Secondary Outcome: Number and Percentage of Participants With Best Overall Response With Partial or Complete Response
Description: Frequency (%) of response-evaluable patients with best overall response of partial or complete response as determined by revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline (version 1.1).
Time Frame: Up to 1 year
Population: Patients with complete response or partial response among response-evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion | Part B, Neuroblastoma | Part C, Medulloblastoma/CNS PNET | Part D, Rhabdomyosarcoma
Number analyzed (Participants) | 4 | 5 | 4 | 9 | 8 | 6 | 19 | 10 | 10
Participants | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0

8. Secondary Outcome: Mean Fold Change in Gamma H2AX in Peripheral Blood Mono Nuclear Cells
Description: Mean (SD) of the increase in gamma H2AX at 4 hours versus baseline among patients in Part A stratified by dose level.
Time Frame: Up to 1 day
Population: Part A patients with data available. Per study protocol, pharmacodynamics were not required for Parts B, C, or D, therefore, data were not collected and will not be collected.
Measure: Mean (Standard Deviation); unit: Fold change
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5
Number analyzed (Participants) | 3 | 3 | 2 | 3 | 3
Fold change | 4.5 (4.18) | 0.45 (0.24) | 3.78 (0.72) | 2 (2.17) | 10 (11.89)

9. Secondary Outcome: Number and Percentage of Part B Neuroblastoma Participants With MYCN Amplification
Description: Frequency (%) of Part B Neuroblastoma participants with MYCN amplification.
Time Frame: Assessed at Baseline
Population: Only Part B eligible patients. Per study protocol, data for Parts A, C, and D were not and will not ever be collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B, Neuroblastoma
Number analyzed (Participants) | 19
Participants | 2

ADVERSE EVENTS:
Time Frame: Up to 12 months
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. Ineligible patients are excluded from reporting of adverse events. All-Cause Mortality includes all deaths collected on the study.
Arm/Group | Part A, Dose Level 1 | Part A, Dose Level 2 | Part A, Dose Level 3 | Part A, Dose Level 4 | Part A, Dose Level 5 | Part A, PK Expansion | Part B, Neuroblastoma | Part C, Medulloblastoma/CNS PNET | Part D, Rhabdomyosarcoma
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/5 | 0/4 | 0/10 | 0/8 | 0/6 | 1/19 | 1/10 | 1/10
Serious Adverse Events (participants affected / at risk) | 4/4 | 2/5 | 3/4 | 10/10 | 6/8 | 6/6 | 11/19 | 9/10 | 7/10
Other Adverse Events (participants affected / at risk) | 4/4 | 5/5 | 4/4 | 10/10 | 8/8 | 6/6 | 19/19 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Dose Level 1 (N=4) | Part A, Dose Level 2 (N=5) | Part A, Dose Level 3 (N=4) | Part A, Dose Level 4 (N=10) | Part A, Dose Level 5 (N=8) | Part A, PK Expansion (N=6) | Part B, Neuroblastoma (N=19) | Part C, Medulloblastoma/CNS PNET (N=10) | Part D, Rhabdomyosarcoma (N=10)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 1 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fever (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 4 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 3 | 1 | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Infections and infestations - Other, CMV VIREMIA (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other, Retropharyngeal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 2 | 1 | 7 | 1 | 2 | 5 | 2 | 1
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, PROGRESSIVE DISEASE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, TUMOR DEBULKING FOR RAP (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 0 | 2 | 5 | 2 | 1 | 6 | 6 | 3
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Optic nerve disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0 | 5 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, BRADYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, UPPER AIRWAY OBSTRUCTION -BULBAR IN NATURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, TUMOR BLEEDING (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Surgical and medical procedures - Other, BILATERAL LUNG WEDGE RESECTIONS (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, CYST DECOMPRESSION SURGERY (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, VENTRICULOPERITONEAL SHUNT (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2
Weight gain (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 1 | 0 | 1 | 3 | 1 | 1 | 3 | 3 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A, Dose Level 1 (N=4) | Part A, Dose Level 2 (N=5) | Part A, Dose Level 3 (N=4) | Part A, Dose Level 4 (N=10) | Part A, Dose Level 5 (N=8) | Part A, PK Expansion (N=6) | Part B, Neuroblastoma (N=19) | Part C, Medulloblastoma/CNS PNET (N=10) | Part D, Rhabdomyosarcoma (N=10)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4 | 3 | 5 | 4 | 2 | 3 | 4 | 7
Abducens nerve disorder (Nervous system disorders) | 0 | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 1 | 4 | 4 | 2 | 10 | 8 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 2 | 3 | 1 | 2 | 4 | 3 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 4 | 5 | 6 | 1 | 2 | 4 | 3
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 4 | 3 | 2 | 9 | 6 | 3 | 14 | 8 | 7
Anorexia (Metabolism and nutrition disorders) | 3 | 2 | 3 | 4 | 5 | 4 | 3 | 5 | 6
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 3 | 1 | 3 | 1 | 3 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 1 | 2 | 5 | 1 | 10 | 7 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 2
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 5 | 2 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood and lymphatic system disorders - Other, (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood and lymphatic system disorders - Other, SPLENOMEGALY (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 1 | 3 | 0 | 1
Blurred vision (Eye disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 1
Cholesterol high (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Concentration impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Congenital, familial and genetic disorders - Other, CONGENITAL HEART DISEASE (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 3 | 0 | 2 | 0 | 4 | 2 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 6 | 3 | 0 | 6 | 2 | 5
Creatinine increased (Investigations) | 1 | 1 | 1 | 3 | 2 | 1 | 3 | 3 | 1
Cushingoid (Endocrine disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3 | 3
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 2 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 5 | 3 | 8 | 6 | 5 | 11 | 7 | 7
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 2 | 2 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 1 | 2 | 2 | 0 | 1 | 0 | 1 | 0
Dysesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1
Dysmenorrhea (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 4
Ear and labyrinth disorders - Other, (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear and labyrinth disorders - Other, EUSTACHIAN TUBE OBSTRUCTION (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Edema face (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Endocrine disorders - Other, (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 1 | 0 | 1 | 4 | 0
Esophageal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
External ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Eye disorders - Other, ERYTHEMA (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, EYE TWITCH (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, MYOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Eye disorders - Other, OCULAR DISCHARGE (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye disorders - Other, Visual disturbance (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Facial muscle weakness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial nerve disorder (Nervous system disorders) | 0 | 2 | 2 | 3 | 0 | 0 | 0 | 3 | 0
Facial pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Fatigue (General disorders) | 3 | 2 | 4 | 6 | 6 | 4 | 8 | 7 | 8
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 0 | 3 | 2 | 0 | 5 | 0 | 5
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
GGT increased (Investigations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 2 | 1 | 3 | 1 | 1 | 0 | 2 | 2
Gastric hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0
Gastrointestinal disorders - Other, CHIPPED TEETH (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, ERUCTATION (BELCHING) (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, HEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, PRESUMED FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorders - Other, RECTAL FISSURE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal disorders - Other, THRUSH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other, GENERALIZED EDEMA (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
General disorders and administration site conditions - Other, Mild itching on Arms and legs (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
General disorders and administration site conditions - Other, SEASONAL ALLERGIES (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Glossopharyngeal nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Growth hormone abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 2 | 2 | 5 | 6 | 3 | 4 | 6 | 4
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 1
Hematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 0 | 2
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 5 | 5 | 1 | 4 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 3 | 1 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 2 | 2 | 1 | 5 | 3 | 3
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Hypersomnia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 3 | 3 | 3 | 2 | 0 | 3
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 4 | 2 | 2 | 6 | 3 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1 | 5 | 1 | 3 | 5 | 3
Hypoglossal nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 5 | 5 | 1 | 4 | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4 | 3 | 0 | 3 | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 5 | 2 | 0 | 2 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 6 | 3 | 1 | 5 | 5 | 2
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 2
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0 | 2 | 1 | 4 | 5 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
INR increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Immune system disorders - Other, ASTHMA (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infections and infestations - Other, C. DIFF INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, E COLI (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, E. COLI (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, FLU (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infections and infestations - Other, HUMAN RHINOVIRUS/ENTEROVIRUS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infections and infestations - Other, STAPHYLOCOCUS AUREUS ON TRACHEAL ASPIRATE (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infusion site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3
Intracranial hemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ABSOLUTE NEUTROPHIL COUNT INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, ALK PHOS DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ALKALINE PHOSPHATASE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, ANION GAP ELEVATED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Investigations - Other, ANION GAP INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, AST DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, BICARBONATE DECREASE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, BICARBONATE DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, BICARBONATE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, BICARBONATE SERUM LOW (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Investigations - Other, BUN DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, BUN ELEVATED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Investigations - Other, BUN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, BUN increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, CO2 DECREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, CRP INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, DECREASED BUN (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED BUN (Investigations) | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED CHLORIDE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, ELEVATED CO2 (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, ELEVATED LDH (Investigations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Investigations - Other, FERRITIN INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, FSH Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, HYPERCHLOREMIA (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, HYPOCHLOREMIA (Investigations) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, INCREASED NEUTROPHIL COUNT (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, INCREASED WBC (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, LOW CREATININE (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, PAPULE (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, PT ELEVATED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, SED RATE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Investigations - Other, SERUM PHOSPHORUS ELEVATED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, TOTAL PROTEIN DECREASED (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Investigations - Other, VIT D DEFICIENCY (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, WHITE BLOOD CELL INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Investigations - Other, bicarbonate serum low (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Investigations - Other, elevated LDH (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irregular menstruation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3 | 1
Lip infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Localized edema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lordosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 4 | 4 | 4 | 8 | 5 | 4 | 12 | 8 | 8
Malaise (General disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolism and nutrition disorders - Other, CACHEXIA (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Metabolism and nutrition disorders - Other, CUSHINGOID SYNDROME (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metabolism and nutrition disorders - Other, Hyperalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Metabolism and nutrition disorders - Other, VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, ANKLE PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, GROWTH PLATE ABNORMALITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, KYPHOSCOLIOSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, OPHTHALMOPLEGIA LEFT (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, RESTLESS LEGS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 1 | 2
Nail discoloration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 5 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 5 | 5 | 4 | 12 | 8 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Nervous system disorders - Other, (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, ABDUCENS NEUROPATHY - BILATERAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, ALTERED MENTAL STATUS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, CEREBELLAR DYSFUNCTION (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, COGNITIVE IMPAIRMENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, DECREASED DTRS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, DIPLOPIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, DYSMETRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, EXOTROPIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, FACIAL NERVE PALSY LEFT (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, HORNER'S SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nervous system disorders - Other, HYPOTROPIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, LEFT SIDED FACIAL TWITCHING (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, MILD DYSMETRIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, NYSTAGMUS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, PARASOMNIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nervous system disorders - Other, RIGHT SIDED HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, SEIZURE DISORDER (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervous system disorders - Other, SLIGHT NYSTAGMUS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nervous system disorders - Other, TRANSIENT NEUROLOGICAL SYMPTOMS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nervous system disorders - Other, VENTRICULOMEGALY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1 | 6 | 2 | 1 | 10 | 5 | 4
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 2 | 0
Nystagmus (Nervous system disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0
Oculomotor nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1
Olfactory nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pain (General disorders) | 0 | 0 | 0 | 2 | 2 | 1 | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 5 | 1 | 0 | 4 | 2 | 3
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Papilledema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1 | 1 | 1 | 0 | 3 | 0 | 1 | 2
Personality change (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Platelet count decreased (Investigations) | 3 | 2 | 1 | 7 | 4 | 2 | 12 | 6 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 5
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Psychiatric disorders - Other, (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Psychiatric disorders - Other, PTSD & ATTACHMENT DISORDER (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rectal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal and urinary disorders - Other, GLUCOSURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, GLUCOSURIA G1 (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, KETONURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, NOCTURNAL ENURESIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, BRADYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, DECREASED BREATH SOUNDS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, SEASONAL ALLERGIES (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 2 | 0
Serum amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 2 | 4 | 3 | 2 | 2 | 2 | 5
Skin and subcutaneous tissue disorders - Other, (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ECCHYMOSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, ERYTHMATOUS RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, HAIR DEPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, HAIR HYPOPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, LINEAR STRIAE (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Laceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Lip Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, MACULAR RASH (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, Nail Dystrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PALLOR (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PERINEAL SKIN BREAKDOWN (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, PETECHIAL RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SKIN TEAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin and subcutaneous tissue disorders - Other, SMEGMA (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, TUMOR BLEEDING (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, Toxic Erythema of Chemotherapy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Social circumstances - Other, (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 2 | 2 | 1 | 1
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0
Stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, G-tube placement (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 5 | 3 | 8 | 6 | 3 | 13 | 10 | 8
Watering eyes (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight gain (Investigations) | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 0 | 1 | 2 | 2 | 2 | 0 | 3 | 4 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
White blood cell decreased (Investigations) | 3 | 2 | 2 | 8 | 5 | 4 | 12 | 6 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/32/NCT02095132/Prot_SAP_001.pdf